CLINICAL TRIAL: NCT05225116
Title: Safety and Efficacy of Lenvatinib and Anti-PD1 Antibody Combined With Radiotherapy Neoadjuvant Treatment for Resectable Hepatocellular Carcinoma With PVTT,Prospective, Multicenter, Single-arm Study
Brief Title: Safety and Efficacy of Lenvatinib and Anti-PD1 Antibody Combined With Radiotherapy Neoadjuvant Treatment for Resectable Hepatocellular Carcinoma With PVTT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21323-0-03
Record Dates: First submitted 2022-01-23; First posted 2022-02-04 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; lenvatinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Lenvatinib+Radiotherapy (Experimental)
  Interventions: Drug: Sintilimab; Drug: Lenvatinib; Radiation: radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be at a dose of 200mg,Q3W
Drug: Lenvatinib — On the first day of the trial, Lenvatinib will be taken orally once daily （8mg/day ≤ 60kg or 12mg/day ≥60kg).
Radiation: radiotherapy — Radiotherapy will be completed within two weeks at a dose of 300cGy× 10 fraction

SUMMARY:
Patients with hepatocellular carcinoma with PVTT can benefit from surgical resection and radiotherapy. As the rapid development of systematic treatment in hepatocellular carcinoma, ICIs neoadjuvant therapy is being actively explored .But there is no evidence to prove the safety and efficacy of lenvatinib and anti-PD1 antibody combined with radiotherapy neoadjuvant treatment for resectable hepatocellular carcinoma with PVTT. This study intends to supplement the evidence of benefit in such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70, with no gender limitation;
2. HCC patients who strictly met the clinical diagnostic criteria of The Code for The Diagnosis and Treatment of Primary Liver Cancer (2019 edition) or were confirmed by histopathological or cytological examination;
3. BCLC stage C, no distant metastasis;
4. Patients with PVTT of type VP1-2-3-4 according to Japanese VP Classification;
5. The primary tumor can be resected (the remaining liver has complete vascular structure and sufficient liver volume, in line with the decision-making system of safe liver resection)
6. ECOG score 0-1;
7. Child-Pugh score ≤7;
8. If the patient is HBV antigen positive, HBV DNA < 500 IU/ mL, conventional antiviral treatment;
9. The major organs meeting the following criteria:

   1. Adequate bone marrow function, defined as: Absolute neutrophil count (ANC ≥ or equal to 1.5 X 10 ^ 9 per liter (/ L)) Hemoglobin (Hb ≥ 8.5 g/dL) Platelet count ≥ 75×10 ^ 9 / L.
   2. Adequate liver function, defined as: Albumin > 2.8 g/dL Bilirubin is 3.0 mg/dL or less Aspartate aminotransferase (AST), alkaline phosphatase (ALP) and alanine aminotransferase (ALT) are less than or equal to 5 ULN.
   3. Adequate coagulation function, defined as an international standardized ratio ( (INR) of 2.3 or less.
   4. Adequate renal function was defined as creatinine clearance greater than 40 mL/min (mL/min), calculated according to the Cockcroft and Gault formulas.
   5. Adequate pancreatic function, defined as amylase and lipase. = 1.5 x ULN.
10. Adequate control of blood pressure (BP) with up to 3 antihypertensive drugs, defined as BP-lt at screening time; = 150/90 mmHg (mmHg), and there was no change in antihypertensive therapy 1 week prior to cycle 1 / day 1.
11. Patients are expected to survive longer than 3 months.
12. No pregnancy or pregnancy plan.
13. Subjects voluntarily joined the study and signed informed consent with good compliance and follow-up.

Exclusion Criteria:

1. Extrahepatic metastasis of primary hepatocellular carcinoma;
2. Diffuse liver cancer;
3. Patients who had previously received targeted drugs or immune checkpoint inhibitors;
4. allergic to Lenvatinib or PD-1 inhibitor ingredients;
5. Patients with grade II or higher myocardial ischemia or myocardial infarction and poorly controlled arrhythmias (including QTc interval ≥470 ms); Patients with grade III ~ IV cardiac insufficiency according to NYHA standard, or left ventricular ejection fraction (LVEF) < 50% as indicated by color doppler echocardiography;
6. abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds or APTT > 1.5ULN), with bleeding tendency or receiving thrombolytic or anticoagulant therapy;
7. pregnant or breast-feeding women; Fertile patients unwilling or unable to take effective contraceptive measures;
8. have a history of mental illness or abuse of psychotropic drugs;
9. patients with co-HIV infection;
10. a history of liver resection, liver transplantation, interventional therapy, and other malignant tumors;
11. patients with active infection;
12. contraindications to radiotherapy;
13. Patients with poor compliance such as floating population;
14. participants in clinical trials of other experimental drugs or devices within 4 weeks;
15. those considered unsuitable for inclusion by the researcher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Safety(CTCAE v5.0) | up to 5 years
  Number of patients who reported incidence of grade ≥3 treatment related adverse events.
Number of patients who complete pre-op treatment and proceed to surgery | up to 5 years
  Number of patients who complete pre-op treatment and proceed to surgery

SECONDARY OUTCOMES:
Major Pathological Response(MPR) | Within 3 months after surgery
  Survival tumor ≤10% during surgery
Objective Response Rate(ORR) | within 1 week before surgery
  Efficacy included objective response (includes complete and partial response) according to modified RECIST 1.1 for HCC
Imaging-pathology Concordance Rate | Within 3 months after surgery
  Imaging-pathology Concordance Rate
PVTT regression rate | Within 3 months after surgery
  The fading rate of PVTT
Median Overall survival(mOS) | up to 5 years
  mOS is defined as the median difference (in months) between the date of study enrollment to the date death due to any cause
Recurrence free survival(RFS) | 1 year after surgery
  From radical resection to the date of the first documented tumor into recurrence or death from any cause, whichever occurred first

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li G, Shu B, Zheng Z, Yin H, Zhang C, Xiao Y, Yang Y, Yan Z, Zhang X, Yang S, Li G, Dong J. Safety and efficacy of radiotherapy combined with lenvatinib plus PD-1 inhibitors as neo-adjuvant therapy in hepatocellular carcinoma with portal vein thrombus: protocol of an open-label, single-arm, prospective, multi-center phase I trial. Front Oncol. 2022 Nov 24;12:1051916. doi: 10.3389/fonc.2022.1051916. eCollection 2022. PMID 36505833